CLINICAL TRIAL: NCT06565325
Title: The Immediate Effect of Combined Terminal Knee Extension Exercise With Audible Cues on Vastus Medialis Muscle Motor Unit Behavior in Healthy Individuals
Brief Title: The Immediate Effect of Combined Terminal Knee Extension Exercise With Audible Cues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Komsak Sinsurin, Asst.Prof.Dr., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-CIRB 2024/021.0802
Record Dates: First submitted 2024-08-11; First posted 2024-08-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Muscle Weakness
Keywords: Terminal Knee Extension Exercise; Audible Cues; Therapeutic exercise; Muscle strength
MeSH Terms: conditions — Muscle Weakness | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There are 2 groups in the current study including exercise with and without audible cues.
Who Masked: Participant
Masking Description: Participant group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Terminal Knee Extension Exercise with Audible Cues
  Interventions: Behavioral: Exercise + Audible Cues
- Control group (Active Comparator): Terminal Knee Extension Exercise without Audible Cues
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise + Audible Cues — Combined Terminal Knee Extension Exercise with Audible Cues
  Other Names: Metronome
  Arms: Experimental group
Behavioral: Exercise — Terminal Knee Extension Exercise
  Arms: Control group

SUMMARY:
Typically, patients perform TKE by themselves after exercise prescription. The investigators thought that a lack of attention and preferred speed of patients might not provide the best outcome. Therefore, an increased effectiveness of TKE is interesting for physical therapy implication. Besides, adding sensory input which is audible cues or rhythm during exercise may enhance the efficacy of the exercise by increasing neuromuscular control and function.

Therefore, the study aimed to investigate the immediate effects of combined TKE with audible cues on motor unit behavior. The researchers expect that adding rhythm from the metronome will enhance neuromuscular control which may change motor unit behavior of VM muscle. The findings of the study may have helped explain the mechanism behind the acute effects of combined TKE with audible cues on VM function and their potential application in the field of physical therapy.

This study aims to investigate the immediate effect of combined TKE with audible cues on motor unit behavior in healthy participants and to investigate reliability of decomposition electromyography procedure during single leg squat.

DETAILED DESCRIPTION:
A metronome will be used to provide rhythmic exercise. Participants will stand with their feet in line with their shoulders as starting position and straping at the knee. Exercise intensity is 60% of the 1RM weight. At the beginning of the exercise, participants will be asked to bend their knees following the pull of the resistance and exert force to straighten the knee (10 times/set and 3 sets). 180 seconds of resting will be allowed between sets.

ELIGIBILITY:
Inclusion Criteria:

* Aged range between 18 and 30 years
* BMI of 18.5-25 kg/m2
* Male or female
* Lightly active or sedentary {Physical activity level (PAL= 1.4-1.69)}

Exclusion Criteria:

* History of serious injury or operation of lower back and lower extremities such as fracture
* Musculoskeletal problems of lower back and lower extremities in 6 months before the study
* Single-leg stance test < 43 seconds (26). and range of weight-bearing lunge test < 9.1 cm

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Motor unit firing rate | At the end of Cycle 1 (each cycle is 1 day)
  one parameter to explain the motor unit behavior of vastus medialis muscle
Peak motor action potential | At the end of Cycle 1 (each cycle is 1 day)
  one parameter to explain the motor unit behavior of vastus medialis muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Nakhon Pathom, Salaya, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suntornon P, Kiratisin P, Sinsurin K, Nitkotom S, Sonsukong A, Thong-On S, Watcharakeunkhan P, Sakunkaruna T. Exercise synchronized with audible cues preserves motor unit action potential: a randomized control trial study. BMC Sports Sci Med Rehabil. 2025 Dec 17. doi: 10.1186/s13102-025-01490-y. Online ahead of print. PMID 41402906